CLINICAL TRIAL: NCT01199471
Title: A Multi-center Registry to Estimate the Behavior of Chinese Anesthesiologists Practicing General Anesthesia With Sevoflurane
Brief Title: Estimate the Behavior of Chinese Anesthesiologists Practicing General Anesthesia With Sevoflurane
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Collaborators: Rundo-Cronova International Pharmaceuticals Research & Development Co., Ltd. (Unknown)
Responsible Party: Sponsor
Other Study IDs: P12-563
Record Dates: First submitted 2010-08-31; First posted 2010-09-13 (Estimated); Results first posted 2012-01-06 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Anesthesia, General
Keywords: Sevoflurane; Physician's Practice Patterns; Economics, Pharmaceutical; Chinese

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Chinese Patients Requiring Surgery with Anesthesia: Chinese patients 18 to 70 years of age, meeting the American Society of Anesthesiologists (ASA) Physical Status Class 1 (normal healthy), Class 2 (mild systemic disease), or Class 3 (severe systemic disease), who underwent surgery requiring general anesthesia (sevoflurane) administered per local Prescribing Information and endotracheal intubation or laryngeal mask airway (LMA).

SUMMARY:
This registry is primarily aiming to demonstrate the correlation between good practices of anesthesiologists and patient related outcomes including decreased overall anesthesia cost. The investigators would also like to demonstrate how the training background, and experience in inhalational anesthesia of the anesthesiologist influence their daily practice. At the end of the registry, the investigators would be able to demonstrate the influence of different practice pattern on patient related outcomes between the sites at which anesthesiologists follow modern anesthesiology practice based on their training/experience background and at which anesthesiologists do not follow same type of practice due to lack of their inhalational anesthesia training/experience.

ELIGIBILITY:
Inclusion Criteria:

1. ASA (American Society of Anesthesiologists) physical status (a requirement of the patient's physical status): I to III
2. Age from 18 to 70 years
3. Surgery requiring general anesthesia with endotracheal intubation or laryngeal mask airway.

Exclusion Criteria:

1. History of significant cardiovascular, pulmonary, renal, hepatic or central nervous system disease or muscle disease.
2. Hypersensitivity or unusual response to any halogenated anesthetics.
3. Personal or familial history of malignant hyperthermia.
4. Female patients either pregnant or breast feeding.
5. General anesthesia is administered with total intravenous anesthesia (TIVA) of propofol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese patients undergoing surgery requiring general anesthesia with endotracheal intubation or laryngeal mask airway
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2010-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yue Kang, MD, Study Director — Abbott
Locations (40):
- China (40):
  - Site Reference ID/Investigator# 43073, Guangzhou, Guangdong
  - Site Reference ID/Investigator# 43072, Guangzhou, Guangdong
  - Site Reference ID/Investigator# 46407, Guangzhou, Guangdong
  - Site Reference ID/Investigator# 43076, Guangzhou, Guangdong
  - Site Reference ID/Investigator# 43077, Guangzhou, Guangdong
  - Site Reference ID/Investigator# 43066, Harbin, Heilongjiang
  - Site Reference ID/Investigator# 43068, Harbin, Heilongjiang
  - Site Reference ID/Investigator# 43071, Wuhan, Hubei
  - Site Reference ID/Investigator# 43070, Wuhan, Hubei
  - Site Reference ID/Investigator# 43065, Chengdu, Sichuan
  - Site Reference ID/Investigator# 43064, Chengdu, Sichuan
  - Site Reference ID/Investigator# 43056, Beijing
  - Site Reference ID/Investigator# 43060, Beijing
  - Site Reference ID/Investigator# 46406, Beijing
  - Site Reference ID/Investigator# 43058, Beijing
  - Site Reference ID/Investigator# 44382, Beijing
  - Site Reference ID/Investigator# 43059, Beijing
  - Site Reference ID/Investigator# 43062, Beijing
  - Site Reference ID/Investigator# 43063, Beijing
  - Site Reference ID/Investigator# 43061, Beijing
  - Site Reference ID/Investigator# 43057, Beining
  - Site Reference ID/Investigator# 44384, Daqing
  - Site Reference ID/Investigator# 44383, Guangzhou
  - Site Reference ID/Investigator# 43074, Guangzhou
  - Site Reference ID/Investigator# 43067, Harbin
  - Site Reference ID/Investigator# 43051, Jiangsu
  - Site Reference ID/Investigator# 43015, Shanghai
  - Site Reference ID/Investigator# 43017, Shanghai
  - Site Reference ID/Investigator# 41554, Shanghai
  - Site Reference ID/Investigator# 46405, Shanghai
  - Site Reference ID/Investigator# 43012, Shanghai
  - Site Reference ID/Investigator# 43014, Shanghai
  - Site Reference ID/Investigator# 43011, Shanghai
  - Site Reference ID/Investigator# 43018, Shanghai
  - Site Reference ID/Investigator# 46404, Shanghai
  - Site Reference ID/Investigator# 43069, Wuhan, Hubei
  - Site Reference ID/Investigator# 43052, Zhejiang
  - Site Reference ID/Investigator# 43053, Zhejiang
  - Site Reference ID/Investigator# 43054, Zhejiang
  - Site Reference ID/Investigator# 43055, Zhejiang

RESULTS

PARTICIPANT FLOW:
Groups:
- Chinese Patients Requiring Surgery With Anesthesia: Chinese patients 18 to 70 years of age, meeting the American Society of Anesthesiologists (ASA) Physical Status Class 1 (normal healthy), Class 2 (mild systemic disease), or Class 3 (severe systemic disease), who underwent surgery requiring general anesthesia administered per the local Prescribing Information and endotracheal intubation or laryngeal mask airway (LMA). Note, 3 patients were excluded from all analyses who did not meet ASA Physical Status Class 1 through 3.
Period: Overall Study
Arm/Group | Chinese Patients Requiring Surgery With Anesthesia
Started | 4000 (3 patients who did not meet ASA Physical Status Class 1 - 3 were excluded from all analyses.)
Completed | 3994
Not Completed | 6
Not completed — Protocol Violation | 4
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Chinese Patients Requiring Surgery With Anesthesia
Number analyzed (Participants) | 3997
Age Continuous [Median (Inter-Quartile Range); unit: years] | 46 [35 to 56]
Age Continuous [Mean (Standard Deviation); unit: years] | 45.26 (13.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2344
  Male | 1653
Region of Enrollment [Number; unit: participants]
  China | 3997

OUTCOME MEASURES:

1. Primary Outcome: Anesthesiologist Satisfaction With the Anesthesia Recorded at the End of the Operation Using a Numeric Analog Scale (NAS)
Description: Anesthesiologist satisfaction with the anesthesia administered to each patient during surgery was recorded at the end of the operation using a Numeric Analog Scale (NAS) from 0 (not satisfied at all) to 10 (completely satisfied) are summarized.
Time Frame: Within 24 hours
Population: 400 participating anesthesiologists evaluated their satisfaction with anesthesia (sevoflurane) administered to patients during surgery. All available data for 3,993 patients are included and summarized.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Chinese Patients Requiring Surgery With Anesthesia: Chinese patients 18 to 70 years of age, meeting the American Society of Anesthesiologists (ASA) Physical Status Class 1 through 3, who underwent surgery requiring general anesthesia administered per the local Prescribing Information and endotracheal intubation or laryngeal mask airway (LMA).
Arm/Group | Chinese Patients Requiring Surgery With Anesthesia
Number analyzed (Participants) | 3993
units on a scale | 8.85 (0.96)

2. Primary Outcome: Patient Satisfaction With the Anesthesia Recorded at the End of the Operation Using a Numeric Analog Scale (NAS)
Description: Patient satisfaction with the anesthesia recorded at the end of the operation within 24 hours using a numeric analog scale (NAS) from 0 (not satisfied at all) to 10 (completely satisfied) are summarized.
Time Frame: Within 24 hours
Population: All available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chinese Patients Requiring Surgery With Anesthesia
Number analyzed (Participants) | 3972
units on a scale | 8.88 (0.93)

3. Secondary Outcome: Time to Loss of Consciousness of Patients Administered Anesthesia
Description: The time to loss of consciousness was measured from commencement of administration of anesthesia to the patient's loss of consciousness (no response to command).
Time Frame: Up to 10 minutes
Population: All available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Chinese Patients Requiring Surgery With Anesthesia
Number analyzed (Participants) | 3921
minutes | 1.65 (0.92)

4. Secondary Outcome: Time to Intubation of Patients
Description: The time to intubation of the patients was measured from the commencement of administration of anesthesia to intubation of each patient.
Time Frame: Up to 10 minutes
Population: All available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Chinese Patients Requiring Surgery With Anesthesia
Number analyzed (Participants) | 3944
minutes | 4.06 (1.74)

5. Secondary Outcome: Time to Eye Opening of Patients
Description: Time to eye opening of patients was measured by the time from cessation of anesthesia administration to opening of the patients' eyes. After cessation of anesthesia, the investigators lightly tapped on the patients forehead or shoulder and asked the patients to open their eyes. This process was repeated about every minute until the patients opened their eyes.
Time Frame: Every minute after cessation of anesthesia until the patient opened his/her eyes
Population: All available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Chinese Patients Requiring Surgery With Anesthesia
Number analyzed (Participants) | 2605
minutes | 14.02 (8.35)

6. Secondary Outcome: Time to Extubation of Patients
Description: The time to extubation of patients was measured from cessation of anesthesia administration to tracheal extubation of the patient.
Time Frame: Every minute after cessation of anesthesia until the patient was extubated
Population: All available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Chinese Patients Requiring Surgery With Anesthesia
Number analyzed (Participants) | 2617
minutes | 16.33 (9.59)

ADVERSE EVENTS:
Time Frame: All adverse events experienced by patients that occurred during the course of the study were reported. Adverse events occurring during the study were reported up to 30 days after the last dose of study treatment.
Arm/Group | Chinese Patients Requiring Surgery With Anesthesia
Serious Adverse Events (participants affected / at risk) | 0/3997
Other Adverse Events (participants affected / at risk) | 43/3997
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chinese Patients Requiring Surgery With Anesthesia (N=3997)
Arrhythmia (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 4 (4)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Postoperative nausea and vomiting (Gastrointestinal disorders) | 6 (6)
Allergic reaction (Immune system disorders) | 1 (1)
Asthma (Immune system disorders) | 1 (1)
Slow heart rhythm (Investigations) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 14 (14)
Hypertension (Vascular disorders) | 7 (8)
Agitation during the operation (Nervous system disorders) | 2 (2)
Emergence agitation (Nervous system disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Types of surgery not restricted/stratified in the study and no standard practice in China on inhalation and intravenous anesthesia methods may skew/bias results. Gaps in study design and multiple outcome parameters make drawing conclusions difficult.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.